CLINICAL TRIAL: NCT03841448
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study of Cemdisiran in Adult Patients With IgA Nephropathy
Brief Title: A Study of Cemdisiran in Adults With Immunoglobulin A Nephropathy (IgAN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early having identified clinically meaningful magnitude of proteinuria reduction due to cemdisiran (study goal). Participants completed DBT period&were in OLE period. Sponsor had no concerns with safety&integrity of participants.
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-CC5-005; 2018-002716-27 (EudraCT Number)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: IgA Nephropathy (IgAN); Berger Disease; Glomerulonephritis, IgA
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind Treatment (DBT) Period: Cemdisiran (Experimental): Participants received cemdisiran, 600 milligrams (mg), subcutaneous (SC) injection, once every 4 weeks (Q4W) in combination with standard of care treatment up to a maximum of 38 weeks in the DBT period.
  Interventions: Drug: Cemdisiran
- DBT Period: Placebo (Placebo Comparator): Participants received cemdisiran matching placebo, SC injection, Q4W in combination with standard of care treatment up to a maximum of 38 weeks in the DBT period.
  Interventions: Drug: Placebo
- DBT Period: Cemdisiran to Open-Label Extension (OLE) Period: Cemdisiran (Experimental): Participants who were randomized to receive cemdisiran in the DBT period continued receiving cemdisiran, 600 mg, SC injection, Q4W in combination with standard of care treatment up to a maximum of 88 weeks in the OLE treatment period.
  Interventions: Drug: Cemdisiran
- DBT Period: Placebo to OLE Period: Cemdisiran (Placebo Comparator): Participants who were randomized to receive cemdisiran matching placebo in the DBT period started receiving cemdisiran, 600 mg, SC injection, Q4W in combination with standard of care treatment up to a maximum of 88 weeks in the OLE treatment period.
  Interventions: Drug: Cemdisiran

INTERVENTIONS:
Drug: Placebo — Normal saline (0.9% NaCl) matching volume of cemdisiran doses were administered SC.
  Arms: DBT Period: Placebo
Drug: Cemdisiran — Cemdisiran was administered by SC injection.
  Other Names: ALN-CC5
  Arms: DBT Period: Cemdisiran to Open-Label Extension (OLE) Period: Cemdisiran; DBT Period: Placebo to OLE Period: Cemdisiran; Double-Blind Treatment (DBT) Period: Cemdisiran

SUMMARY:
The purpose of this study is to evaluate the effect of cemdisiran on proteinuria in adults with immunoglobulin A nephropathy (IgAN), who excrete >1 gram (gm) of protein per day despite standard of care, which includes treatment with angiotensin-converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB). These participants are at high risk for progression of kidney disease, which can result in end-stage renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary IgAN
* Currently being treated for IgAN with stable, optimal therapy, including an ACE inhibitor or ARB.
* Has urine protein greater than or equal to 1 gram/24-hour
* Has hematuria (blood cells present in urine)

Exclusion Criteria:

* Has renal disease other than IgAN
* Has a diagnosis of rapidly progressive glomerulonephritis
* Has a diagnosis of Henoch-Schonlein Purpura (IgA Vasculitis)
* Has poor kidney function with estimated glomerular filtration rate (eGFR) <30 milliliters per minute per 1.73 meters square (mL/min/1.73 m^2)
* Has known human immunodeficiency virus (HIV) infection, hepatitis C virus (HCV) infection or hepatitis B virus (HBV) infection
* Has on-going high blood pressure
* Treated with systemic corticosteroids for more than 7 days, or other immunosuppressant agents in the past 6 months
* Received an organ transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (17):
- Canada (3):
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Brampton, Ontario
  - Clinical Trial Site, Toronto, Ontario
- France (3):
  - Clinical Trial Site, Grenoble
  - Clinical Trial Site, La Tronche
  - Clinical Trial Site, Mulhouse
- Malaysia (3):
  - Clinical Trial Site, Kuala Lumpur
  - Clinical Trial Site, Kuantan
  - Clinical Trial Site, Serdang
- Clinical Trial Site, Quezon City, Philippines
- Clinical Trial Site, Singapore, Singapore
- Spain (2):
  - Clinical Trial Site, Córdoba
  - Clinical Trial Site, Girona
- Sweden (2):
  - Clinical Trial Site, Huddinge
  - Clinical Trial Site, Uppsala
- Clinical Trial Site, Taichung, Taiwan
- Clinical Trial Site, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 19 investigative centers in Canada, France, Malaysia, Philippines, Singapore, Spain, Sweden, Taiwan, and the United Kingdom from 30 Sept 2019 to 27 June 2023.
Pre-assignment Details: A total of 31 participants were enrolled in this study to receive cemdisiran or placebo. This study has two parts: Double Blind Treatment (DBT) Period and Open-Label Extension (OLE) Period.
Groups:
- DBT Period: Placebo: Participants received cemdisiran matching placebo, subcutaneous (SC) injection, once every 4 weeks (Q4W) in combination with standard of care treatment up to a maximum of 38 weeks in the DBT period.
- DBT Period: Cemdisiran: Participants received cemdisiran, 600 milligrams (mg), SC injection, Q4W in combination with standard of care treatment up to a maximum of 38 weeks in the DBT period.
- DBT Period: Cemdisiran to OLE Period: Cemdisiran: Participants who were randomized to receive cemdisiran in the DBT period continued receiving cemdisiran, 600 mg, SC injection, Q4W in combination with standard of care treatment up to a maximum of 88 weeks in the OLE treatment period.
Period: Double-blind Treatment (DBT) Period
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran | DBT Period: Placebo to OLE Period: Cemdisiran | DBT Period: Cemdisiran to OLE Period: Cemdisiran
Started | 9 | 22 | 0 | 0
Modified Intent-to-treat (mITT) Analysis Set (mITT Analysis Set included all participants who received any amount of study drug and had at least one post baseline 24-hour urine protein/creatinine ratio (UPCR) assessment.) | 9 | 22 | 0 | 0
Completed | 8 | 21 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Period: Open-Label Extension (OLE) Period
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran | DBT Period: Placebo to OLE Period: Cemdisiran | DBT Period: Cemdisiran to OLE Period: Cemdisiran
Started | 0 | 0 | 8 | 20
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 8 | 20
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 3
Not completed — Study termination by Sponsor | 0 | 0 | 4 | 9
Not completed — Other Reason Not Specified | 0 | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received any amount of study drug.
Groups:
- DBT Period: Cemdisiran: Participants received cemdisiran, 600 mg, SC injection, Q4W in combination with standard of care treatment up to a maximum of 38 weeks in the DBT period.
- Total: Total of all reporting groups
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran | Total
Number analyzed (Participants) | 9 | 22 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (10.4) | 40.5 (10.1) | 39.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 3 | 13 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 7 | 18 | 25
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 12 | 16
  White | 4 | 8 | 12
  Other | 0 | 1 | 1
  Not Reported | 1 | 1 | 2
Urine Protein to Creatinine Ratio [Mean (Standard Deviation); unit: g/g] | 1.972 (0.815) | 1.554 (1.032) | 1.676 (0.979)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in UPCR as Measured in 24-hour Urine at Week 32
Description: UPCR is a way of assessing the amount of protein in the urine. The primary analysis for UPCR was performed using Mixed-Effect Model Repeated Measures (MMRM) approach. Geometric mean (GM)ratios were obtained by exponentially back-transforming the arithmetic mean of change in log-transformed 24h UPCR. Standard error of the mean (SEM) was calculated as exponential (mean of change in log-transformed data) * (standard error of change in log-transformed data). Adjusted GM ratio to baseline and 90% confidence interval (CIs) were calculated by exponentially back-transforming the model-based least square (LS) mean and the corresponding 90% CI.
Time Frame: Baseline to Week 32
Population: mITT Analysis Set included all participants who received any amount of study drug and had at least one post baseline 24-hour UPCR assessment. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Standard Error); unit: percent change
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran
Number analyzed (Participants) | 9 | 22
percent change | 1.095 (0.258) | 0.686 (0.098)
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; p = 0.1032, MMRM; Placebo-adjusted GM Percent Change = -37.367, 90% CI 2-sided [-60.951 to 0.460] — Placebo-adjusted GM percent change, 90% CIs were calculated by exponentially back-transforming the model based LS mean difference (cemdisiran - placebo) and the corresponding 90% CI then subtracting by 1

2. Secondary Outcome: Percent Change From Baseline in 24-hour Proteinuria at Week 32
Description: Proteinuria is high levels of protein in the urine. 24-hour proteinuria assessment included 24-hour urine collections to assess total protein excretion per 24 hours. Analysis was performed using the MMRM model. GM ratios were obtained by exponentially back-transforming the arithmetic mean of change in log-transformed 24h urine protein (UP). SEM was calculated as exp (mean of change in log-transformed data) *(standard error of change in log-transformed data). Adjusted GM ratio to baseline and 90% CIs are calculated by exponentially back-transforming the model-based LS Means and the corresponding 90% CI.
Time Frame: Baseline to Week 32
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: percent change
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran
Number analyzed (Participants) | 9 | 22
percent change | 1.051 (0.266) | 0.671 (0.104)
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; p = 0.1432, MMRM; Placebo-adjusted GM Percent Change = -36.167, 90% CI 2-sided [-61.552 to 5.978] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Partial Clinical Remission at Week 32
Description: Partial clinical remission was defined as having UP <1.0 g/24-hours.
Time Frame: Week 32
Population: mITT Analysis Set included all participants who received any amount of study drug and had at least one post baseline 24-hour UPCR assessment.
Measure: Number; unit: percentage of participants
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran
Number analyzed (Participants) | 9 | 22
percentage of participants | 0 | 22.7
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; p = 0.1177, Cochran-Mantel-Haenszel; p-value was based on Cochran-Mantel-Haenszel test stratified by baseline 24-hour UP (≥1.0 g and <2 g/day versus ≥2.0 g/day); Odds Ratio (OR) = 3.01, 90% CI 2-sided [0.43 to 21.27] — Odds ratio was estimated with logit method using a correction of 0.5 in every cell of the 2x2 table that contains a zero
Statistical Analysis 2: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; Difference in Proportions = 0.23, 90% CI 2-sided [-0.13 to 0.42] — Difference in proportions (cemdisiran - placebo) (90% CI) was based on the Wilson score method with continuity correction

4. Secondary Outcome: Percentage of Participants With >50% Reduction in 24-hour Proteinuria at Week 32
Time Frame: Week 32
Population: mITT Analysis Set included all participants who received any amount of study drug and had at least one post baseline 24-hour UPCR assessment. Percentages are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran
Number analyzed (Participants) | 9 | 22
percentage of participants | 0 | 22.7
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; p = 0.1533, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.02, 90% CI 2-sided [0.45 to 20.34] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; Difference in Proportions = 0.23, 90% CI 2-sided [-0.13 to 0.42] — [estimate comment as in outcome 3, analysis 2]

5. Secondary Outcome: Change From Baseline in UPCR as Measured in a Spot Urine at Week 32
Description: UPCR was calculated by dividing the level of protein in a spot urine test by the creatinine level. Analysis was performed using MMRM model. GM ratios were obtained by exponentially back-transforming the arithmetic mean of change in log-transformed spot UPCR. SEM was calculated as exp (mean of change in log-transformed data) *(standard error of change in log-transformed data). Adjusted GM ratio to baseline and 90% CIs are calculated by exponentially back-transforming the model-based LS Means and the corresponding 90% CI.
Time Frame: Baseline to Week 32
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: gram per gram (g/g)
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran
Number analyzed (Participants) | 9 | 22
gram per gram (g/g) | 1.344 (0.139) | 0.729 (0.109)
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Cemdisiran; Test type: Superiority; p = 0.0021, MMRM; Placebo-adjusted GM Percent Change = -45.771, 90% CI 2-sided [-60.093 to -26.309] — Placebo-adjusted GM percent change, 90% CIs were calculated by exponentially back-transforming the model based LS means difference (cemdisiran - placebo) and the corresponding 90% CI then subtracting by 1

6. Secondary Outcome: Number of Participants With Change From Baseline in Hematuria at Week 32
Description: Hematuria is the presence of blood in the urine. Hematuria from spot urine collections was evaluated to assess the effect of cemdisiran on disease course in participants. The degree of hematuria was assessed by microscopic examination of the spun urine sediment (red blood cell (RBC)/ high power field [hpf]) and by urine dipstick.
Time Frame: Baseline to Week 32
Population: mITT Analysis Set included all participants who received any amount of study drug and had at least one post-baseline 24-hour UPCR assessment. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran
Number analyzed (Participants) | 8 | 20
Participants
  Post-Baseline Category: Negative | 0 | 4
  Post-Baseline Category: Small | 2 | 11
  Post-Baseline Category: Moderate | 2 | 4
  Post-Baseline Category: Large | 4 | 1

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 126 weeks
Population: DBT Period: Safety Analysis Set: All participants who received any amount of study drug.
  DBT + OLE and All Cemdisiran: All Cemdisiran Treated Set: All participants who received at least one dose of cemdisiran, including participants who received cemdisiran during the DB Period and participants who first take placebo during the DB Period and switch to cemdisiran during the OLE Period.
Measure: Count of Participants; unit: Participants
Groups:
- DBT Period: Placebo + OLE Period: Cemdisiran: Participants who were randomized to receive cemdisiran matching placebo in the DBT period started receiving cemdisiran, 600 mg, SC injection, Q4W in combination with standard of care treatment up to a maximum of 88 weeks in the OLE treatment period. The data reported for this group is for the OLE Period only, in which all participants were receiving treatment with cemdisiran.
- DBT Period: Cemdisiran + OLE Period: Cemdisiran: Participants who were randomized to receive cemdisiran in the DBT period continued receiving cemdisiran, 600 mg, SC injection, Q4W in combination with standard of care treatment up to a maximum of 88 weeks in the OLE treatment period. The data reported for this group is for the DBT and OLE Periods inclusively, in which all participants were receiving treatment with cemdisiran.
- All Cemdisiran: All participants who received at least one dose of cemdisiran, including participants who received cemdisiran during the DB Period and participants who first received placebo during the DB Period and switched to cemdisiran during the OLE Period.
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran | DBT Period: Placebo + OLE Period: Cemdisiran | DBT Period: Cemdisiran + OLE Period: Cemdisiran | All Cemdisiran
Number analyzed (Participants) | 9 | 22 | 8 | 22 | 30
Participants | 8 | 19 | 8 | 22 | 30

ADVERSE EVENTS:
Time Frame: DBT Period: from the first dose of study drug up to 38 weeks. OLE Period: from Week 38 up to 88 weeks (up to 126 weeks for both periods combined). All Cemdisiran: from the first dose of study drug up to 126 weeks.
Groups:
- DBT Period: Placebo: Participants received cemdisiran matching placebo, SC injection, Q4W in combination with standard of care up to a maximum of 38 weeks in the DBT period.
Arm/Group | DBT Period: Placebo | DBT Period: Cemdisiran | DBT Period: Placebo + OLE Period: Cemdisiran | DBT Period: Cemdisiran + OLE Period: Cemdisiran | All Cemdisiran
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/22 | 0/8 | 1/22 | 2/30
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/22 | 3/8 | 2/22 | 5/30
Other Adverse Events (participants affected / at risk) | 8/9 | 19/22 | 8/8 | 22/22 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | DBT Period: Placebo (N=9) | DBT Period: Cemdisiran (N=22) | DBT Period: Placebo + OLE Period: Cemdisiran (N=8) | DBT Period: Cemdisiran + OLE Period: Cemdisiran (N=22) | All Cemdisiran (N=30)
Cardiopulmonary failure (Cardiac disorders) | 0/0 | 1/1 | 0/1 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBT Period: Placebo (N=9) | DBT Period: Cemdisiran (N=22) | DBT Period: Placebo + OLE Period: Cemdisiran (N=8) | DBT Period: Cemdisiran + OLE Period: Cemdisiran (N=22) | All Cemdisiran (N=30)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 2 | 3
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 2 | 3
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2
COVID-19 (Infections and infestations) | 0 | 2 | 5 | 9 | 14
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Eyelid infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 2
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1 | 3
Influenza (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Injection site bruising (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 2 | 9 | 5 | 9 | 14
Injection site recall reaction (General disorders) | 0 | 2 | 3 | 2 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Keratosis obturans (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 3
Oedema peripheral (General disorders) | 1 | 3 | 1 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 2
Pain (General disorders) | 0 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2
Pyrexia (General disorders) | 1 | 1 | 2 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Suprapubic pain (General disorders) | 0 | 1 | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 3
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 1 | 1 | 2
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 1
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Superinfection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Viral rash (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 1
Urine sodium increased (Investigations) | 0 | 0 | 0 | 1 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03841448/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT03841448/SAP_001.pdf